CLINICAL TRIAL: NCT06206109
Title: Is There a Relationship Between The Common Extensor Tendon Tears and Clinical-Ultrasonographic Changes in Lateral Epicondylitis?
Brief Title: The Effect of Tendon Tears on Lateral Epicondylitis
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Banu Dilek, Assoc Prof, Dokuz Eylul University
Other Study IDs: LEtendontears
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Lateral Epicondylitis; Tennis Elbow; Tendon Tear
Keywords: Lateral Epicondylitis; Tennis Elbow; Extensor Tendon; Tendon Tear; Ultrasonography
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with common extensor tendon tears: the participants who have common extensor tendon tears demonstrated with ultrasonography.
- without common extensor tendon tears: the participants who do not have common extensor tendon tears demonstrated with ultrasonography.

SUMMARY:
Common extensor tendon (CET) tears that can be detected with ultrasonography (US) may be associated with worsening clinical and other ultrasonographic parameters in patients with LE. In this retrospective evaluation of patients with lateral epicondylitis (LE), the effect of common extensor tendon (CET) tears revealed by ultrasonography (US) with demographic, clinical, and other US findings was investigated.

DETAILED DESCRIPTION:
The files of 227 patients with LE who applied to Dokuz Eylül University Faculty of Medicine, Department of Physical Medicine and Rehabilitation Clinic and met the inclusion and exclusion criteria were reviewed retrospectively.

The demographic characteristics of the patients were recorded.

First of all, common extensor tendon tears, if it existed, were demonstrated with ultrasonography. Then, primary and secondary outcome measures were performed.

Maximum tendon thickness measurements (capitellar - radiocapitellar) and the presence of bone abnormality were detected with ultrasonography of the lateral epicondyle region of the humerus.

The VAS was used to assess pain and was evaluated separately for pain at rest (VAS-rest), at night (VAS-night), and during ADL (VAS-ADL).

Force was applied on the lateral epicondyle using a standard pressure algometer (Baseline®) to evaluate the patient's sensitivity to pain. The pressure at which the patient first felt pain and the average value in kg/cm2 (repeated three times) were recorded.

PRTEE consists of two sub-sections (pain and function): the severity of pain in the elbow and functional deficiencies. The Turkish version of the PRTEE questionnaire was used

The hand dynamometer (JAMAR®) was used to assess the hand grip strength. The patient was positioned with sitting, shoulder adduction, elbow 90° flexion, and forearm in a position between supination and pronation. The average value in kilogram-force (repeated three times). Between repeated measures 1-minute resting, periods were given.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65 years
* diagnosis of LE based on clinical parameters and US findings
* duration of symptoms ranging from 2 to 12 weeks
* agreement to participate in the study

Exclusion Criteria:

* LE findings in the other extremity
* has received any treatment for lateral epicondylitis before
* previous elbow surgery
* history of elbow fracture
* upper extremity muscle weakness due to radiculopathy or neuropathy
* the presence of concurrent neurological, rheumatic, psychiatric, or malignant conditions
* pregnancy
* inability to comply with the study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The files of 227 patients with LE who met the inclusion and exclusion criteria were reviewed retrospectively.
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Patient Rated Tennis Elbow Evaluation (PRTEE) | Day 1
  PRTEE consists of two sub-sections (pain and function): the severity of pain in the elbow and functional deficiencies. The Turkish version of the PRTEE questionnaire was used. PRTEE total score will be evaluated between 0-100. A higher score is associated with worse clinical outcome and function.

SECONDARY OUTCOMES:
Maximum tendon thickness measurements (capitellar - radiocapitellar) | Day 1
  Maximum tendon thickness measurements (capitellar - radiocapitellar) were detected with ultrasonography of the lateral epicondyle region of the humerus
Presence of bone abnormality | Day 1
  The presence of bone abnormality were detected with ultrasonography of the lateral epicondyle region of the humerus
Visual Analog Scale (VAS) | All patients were evaluated for one time.
  The VAS was used to assess pain and was evaluated separately for pain at rest (VAS-rest), at night (VAS-night), and during ADL (VAS-ADL). The VAS score will be evaluated between 0-10. A higher score is consistent with more severe pain.
Hand Grip Strength | Day 1
  The hand dynamometer (JAMAR®) was used to assess the hand grip strength. The patient was positioned with sitting, shoulder adduction, elbow 90° flexion, and forearm in a position between supination and pronation. The average value in kilogram-force (repeated three times). Between repeated measures 1-minute resting, periods were given.
Pain Sensitivity | Day 1
  Force was applied on the lateral epicondyle using a standard pressure algometer (Baseline®) to evaluate the patient's sensitivity to pain. The pressure at which the patient first felt pain and the average value in kg/cm2 (repeated three times) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Dilek, Assoc Prof, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)